CLINICAL TRIAL: NCT02424071
Title: The Effect of Premedication With Melatonin on Postoperative Recovery From Bariatric Surgery: a Prospective Randomised Controlled Cohort Study
Brief Title: The Effect of Premedication With Melatonin on Postoperative Recovery From Bariatric Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Haim Berkenstadt, Director of Anesthesia, Sheba medical center, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHEBA-2015-1841-HB-CTIL
Record Dates: First submitted 2015-04-19; First posted 2015-04-22 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Recovery From Bariatric Surgery
Keywords: melatonin's; quality of recovery
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin group (Active Comparator): Patients will receive a pill containing 5mg of melatonin on the evening before the surgery. Patients will receive another pill containing 5mg of melatonin two hours prior to surgery.
  Interventions: Drug: Melatonin
- Placebo group (Placebo Comparator): Patients will receive a pill containing placebo on the evening before the surgery. Patients will receive another pill containing placebo two hours prior to surgery.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Melatonin
  Arms: Melatonin group
Drug: placebo
  Arms: Placebo group

SUMMARY:
Melatonin has sedative, hypnotic and analgesic properties that make it a good premedication agent before anesthesia and surgery.

In this study the investigators intend to randomise 60 patients undergoing bariatric surgery into two groups. The participants will receive either melatonin or placebo on the evening prior to the surgery, and the same agent two hours before the surgery.

The patients recovery from the surgery and anesthesia will be assessed using the Q0R15 questionnaire. The patients will be asked to take the questionnaire once in the pre-operative clinic, again after the second melatonin or placebo pill before entering the operating room, and once more on the first post-operative day.

DETAILED DESCRIPTION:
Melatonin has sedative, hypnotic, analgesic, antiinflammatory, and chronobiologic properties that make it a good premedication agent before anesthesia and surgery. Patients undergoing surgery in our establishment usually receive benzodiazepines as premedicants to reduce anxiety before the surgery. For bariatric patients benzodiazepines are usually avoided due to side effects which could be deleterious in obese patients.

In this study the investigators intend to randomise 60 patients undergoing bariatric surgery into two groups. The participants will receive either melatonin or placebo on the evening prior to the surgery, and the same agent two hours before the surgery.

The patients recovery from the surgery and anesthesia will be assessed using the Q0R15 questionnaire. The patients will be asked to take the questionnaire once in the pre-operative clinic, again after the second melatonin or placebo pill before entering the operating room, and once more on the first post-operative day.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bariatric surgery

Exclusion Criteria:

* Known allergy to melatonin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Quality of recovery after surgery | First post operative day

CONTACTS AND LOCATIONS:
Overall Officials: Haim Berkenstadt, MD, Study Director — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yousaf F, Seet E, Venkatraghavan L, Abrishami A, Chung F. Efficacy and safety of melatonin as an anxiolytic and analgesic in the perioperative period: a qualitative systematic review of randomized trials. Anesthesiology. 2010 Oct;113(4):968-76. doi: 10.1097/ALN.0b013e3181e7d626. PMID 20823763
- [Background] Caumo W, Torres F, Moreira NL Jr, Auzani JA, Monteiro CA, Londero G, Ribeiro DF, Hidalgo MP. The clinical impact of preoperative melatonin on postoperative outcomes in patients undergoing abdominal hysterectomy. Anesth Analg. 2007 Nov;105(5):1263-71, table of contents. doi: 10.1213/01.ane.0000282834.78456.90. PMID 17959953
- [Background] Fitzpatrick R, Davey C, Buxton MJ, Jones DR. Evaluating patient-based outcome measures for use in clinical trials. Health Technol Assess. 1998;2(14):i-iv, 1-74. No abstract available. PMID 9812244
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- See also: Melatonin NIH fact sheet — http://ods.od.nih.gov/factsheets/list-all/